CLINICAL TRIAL: NCT02437188
Title: Preventing Persistent Post-Surgical Pain and Opioid Use In At-Risk Veterans: Effect of ACT
Acronym: PreACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara A Rakel (Other)
Responsible Party: Sponsor-Investigator, Barbara A Rakel, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201603778
Record Dates: First submitted 2015-04-29; First posted 2015-05-07 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Persistent Post-surgical Pain; Acceptance and Commitment Therapy; Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT plus TAU (Experimental): Participants randomized to receive ACT will be scheduled to attend a 1-day training session before their preoperative clinic visit. The intervention will incorporate both experiential learning and didactic content, will include a summary of the main concepts at the end of the day, and a manual of the main concepts will be sent home with participants so they can practice the exercises prior to and after surgery. Participants will also receive an individualized phone call "booster" intervention 2 weeks after surgery to address any issues and reinforce the information that was given during the workshop. This will be done to facilitate the participant's use of the skills during the postoperative period.
  Interventions: Behavioral: ACT (Acceptance and Commitment Therapy)
- TAU (No Intervention): Current pre-surgery treatment includes a nurse-led patient education class covering the post-operative course and what to expect for pain control and recovery. Patients may be taking analgesia (i.e. opioids and/or non-opioids) preoperatively for a chronic pain condition and are prescribed analgesics, sedatives and/ or anxiolytics immediately prior to surgery. Intraoperatively, regional (i.e., spinal and femoral) anesthesia and analgesia is given and patients receive opioids, non-opioids, anticonvulsants and/or anxiolytics during the immediate postoperative period. Other pain treatments may be used, such as cryotherapy, music therapy, relaxation, imagery, etc. Patients are sent home with analgesia (often a combination medication of an opioid and acetaminophen) for breakthrough pain.

INTERVENTIONS:
Behavioral: ACT (Acceptance and Commitment Therapy) — The 1-day training session with ACT proposed for this study is designed to reduce behavioral avoidance and to enhance acceptance-based coping. The intervention includes: 1) Behavioral Change Training (2.5 hours) involving a) teaching patients how to recognize ineffective patterns of behavior and habits, b) exploring and setting life goals and goals related to mental and physical health, and c) promoting effective and committed actions to achieve these goals despite the urge to do otherwise; 2) Acceptance and Mindfulness Training (2.5 hours) emphasizing new ways of managing troubling thoughts, feelings, and physical sensations (e.g., learning how to recognize, and develop cognitive distance from, unhelpful thoughts and learning how to willingly face experiences that cannot be changed.
  Arms: ACT plus TAU

SUMMARY:
A large number of veterans suffer from distress-based conditions, such as anxiety and depression, putting them at high risk of experiencing persistent pain and prolonged opioid use following surgery. These connections are based on strong and consistent evidence from the literature and our preliminary data. The proposed study adds a 1-day workshop of Acceptance and Commitment Therapy (ACT), followed by an individual "booster" session, to treatment as usual (TAU) to reduce veterans' risk of persistent pain and prolonged opioid use following surgery. ACT has been shown to be effective in reducing chronic pain, anxiety and depression.

This pilot study will establish the feasibility and preliminary efficacy of incorporating ACT into treatment as usual (TAU) to preoperatively target distress-based risk factors. Aim 1 is to establish the feasibility of successfully delivering ACT to at-risk veterans before and after surgery. Aim 2 is to test the preliminary efficacy of ACT on the length and/or amount of pain and opioid use after surgery. Veterans who are anxious or depressed before surgery will be randomly assigned to receive ACT plus TAU or TAU. Outcomes between the two groups will be compared. Aim 3 is to see if PROMIS modules, developed by the National Institute of Health, are useful for assessing pain and other symptoms in veterans. Findings from this study will be used to inform the design and implementation of a larger, well controlled, randomized clinical trial that will evaluate the efficacy of ACT plus TAU for at-risk veterans.

This study will take place at the Iowa City VA Health Care System (VAMC). Veterans scheduled for orthopedic or open abdominal surgery in 1 to 3 months who score high for anxiety or depression will be randomly assigned to attend a 1-day ACT workshop preoperatively, with an individualize "booster" session postoperatively, or to have TAU. Veterans who receive ACT and trainers who provide the treatment will be interviewed to identify barriers and facilitators to providing ACT to at-risk veterans before and after surgery. Other primarily outcomes are pain and opioid use after surgery. Factors that may affect these outcomes will also be measured, including anxiety, depression, substance use disorder, post-traumatic stress disorder, and use of other pain meds.

The investigators expect to gain important knowledge about ways to best include ACT as part of routine care for veterans requiring surgery and about the preliminary efficacy of ACT for the prevention of persistent pain and prolonged opioid use following surgery.

DETAILED DESCRIPTION:
A large number of veterans suffer from distress-based conditions, such as anxiety and depression, putting them at risk of experiencing persistent pain and prolonged opioid use following surgery. Preventing these problems (our long term goal) for the thousands of veterans who undergo surgery each year can have a dramatic impact on quality of life and productivity, including positive effects on mood, daily activities, sleep, cognitive functions, social life and decreased risk of suicide (1, 2). In addition to these benefits for individual veterans, prevention of these problems can significantly reduce the estimated billions of dollars associated with veterans' utilization of the healthcare system as well as costs associated with lost work productivity, including unemployment and disability benefits (3).

Building on strong and consistent evidence showing that high anxiety and depression put veterans at risk for persistent pain and prolonged opioid use following surgery (4, 5), this proposal tests the feasibility and preliminary efficacy of implementing a 1-day training session with Acceptance and Commitment Therapy (ACT) in veterans identified to be at-risk prior to surgery. ACT has been shown to significantly lower distress and disability in patients with chronic pain (6-8) and is particularly valuable intervention for the 80% of veterans who experience some level of psychological distress prior to surgery (9) and the 50% of veterans who report they experience pain on a regular basis (10, 11). Current practice does not include psychological interventions specifically aimed at addressing distress-based conditions prior to surgery. This study is a necessary first step in evaluating the efficacy of this novel intervention during a critical juncture in care to benefit veterans and prevent the devastating consequences of persistent pain and prolonged opioid use following surgery.

This project is based on our interdisciplinary team's research on psychological factors predicting persistent pain after total knee replacement (12) and the effect of ACT on depression and pain in depressed migraine sufferers (13). The design of this 1-day workshop was developed based on feedback given by patients who received ACT during co-I Dindo's preliminary study. The rationale for this research is that, once we determine the feasibility and preliminary efficacy of incorporating this 1-day workshop into treatment as usual (TAU) to preoperatively target distress-based risk conditions, findings from this study will be used to inform the design and implementation of a larger, well controlled, randomized clinical trial that will evaluate the efficacy of ACT plus TAU (ACT + TAU) for at-risk veterans. The following specific aims will be achieved:

* Aim #1: The primary aim of this pilot study is to determine the feasibility of successfully delivering a 1-day ACT intervention with at-risk veterans prior to surgery and an individualized "booster" session after surgery. The following aspects of the intervention will be assessed: 1) the number of at-risk veterans who are willing and able to receive the ACT workshops and individual "booster" sessions; 2) veteran identification of barriers and facilitators to receiving the ACT intervention and utilizing the skills taught; 3) trainer identification of barriers and facilitators to providing the ACT intervention with at-risk veterans before and after surgery; and 4) veteran and trainer suggestions about ways to improve the intervention. These aspects will be assessed primarily through guided open-ended interviews after the ACT workshop and 3 months postoperatively.
* Aim #2: To determine if a 1-day preoperative ACT workshop with an individualized "booster" session postoperatively reduces the length and/or amount of pain and opioid use following surgery when compared to treatment as usual (TAU). Participants will be randomized to ACT + TAU or TAU and record pain and opioid use daily after surgery.
* Aim #3: A secondary, exploratory aim is to determine the usability and utility of the Patient Reported Outcomes Measurement Information System (PROMIS) modules for assessing pain and associated symptoms in veterans. We will compare modules to the Brief Pain Inventory (Pain Interference), the State/Trait Anxiety Inventory (Anxiety), and the Patient Health Questionnaire (PHQ)-9 (Depression).

This project has the potential to infuse what is known about effective treatment of chronic pain into the acute care environment to benefit veterans and improve surgical outcomes. It incorporates an interdisciplinary approach to the care of veterans that attends to the psychology of pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Scheduled for orthopedic surgery at the Iowa City VAMC at least 1 month in the future.
* Movement or resting pain ≥ 3 on a 0-10 NRS.
* Score on the Hamilton Anxiety Rating Scale (HAM-A) ≥ 14; OR
* Score on the Hamilton Depression Rating Scale (HAMD) ≥ 17.

Exclusion Criteria:

* Inability to complete study forms because of either mental incapacity or a language barrier;
* Bipolar or psychotic disorder;
* History of brain injury;
* Complication(s) following surgery requiring reoperation or revision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rakel, PhD, Principal Investigator — University of Iowa
Locations (1):
- Iowa City VAMC, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caffo O, Amichetti M, Ferro A, Lucenti A, Valduga F, Galligioni E. Pain and quality of life after surgery for breast cancer. Breast Cancer Res Treat. 2003 Jul;80(1):39-48. doi: 10.1023/A:1024435101619. PMID 12889597
- [Background] Abyholm AS, Hjortdahl P. [The pain takes hold of life. A qualitative study of how patients with chronic back pain experience and cope with their life situation]. Tidsskr Nor Laegeforen. 1999 Apr 30;119(11):1624-9. Norwegian. PMID 10385806
- [Background] Kerns RD, Sellinger J, Goodin BR. Psychological treatment of chronic pain. Annu Rev Clin Psychol. 2011;7:411-34. doi: 10.1146/annurev-clinpsy-090310-120430. PMID 21128783
- [Background] Carroll I, Hah J, Mackey S, Ottestad E, Kong JT, Lahidji S, Tawfik V, Younger J, Curtin C. Perioperative interventions to reduce chronic postsurgical pain. J Reconstr Microsurg. 2013 May;29(4):213-22. doi: 10.1055/s-0032-1329921. Epub 2013 Mar 5. PMID 23463498
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] McCracken LM, Gutierrez-Martinez O. Processes of change in psychological flexibility in an interdisciplinary group-based treatment for chronic pain based on Acceptance and Commitment Therapy. Behav Res Ther. 2011 Apr;49(4):267-74. doi: 10.1016/j.brat.2011.02.004. Epub 2011 Feb 15. PMID 21377652
- [Background] McCracken LM, Velleman SC. Psychological flexibility in adults with chronic pain: a study of acceptance, mindfulness, and values-based action in primary care. Pain. 2010 Jan;148(1):141-147. doi: 10.1016/j.pain.2009.10.034. Epub 2009 Nov 28. PMID 19945795
- [Background] McCracken LM, Vowles KE. A prospective analysis of acceptance of pain and values-based action in patients with chronic pain. Health Psychol. 2008 Mar;27(2):215-20. doi: 10.1037/0278-6133.27.2.215. PMID 18377140
- [Background] Patton CM, Hung M, Lawrence BD, Patel AA, Woodbury AM, Brodke DS, Daubs MD. Psychological distress in a Department of Veterans Affairs spine patient population. Spine J. 2012 Sep;12(9):798-803. doi: 10.1016/j.spinee.2011.10.008. Epub 2011 Nov 16. PMID 22088603
- [Background] Otis JD, Keane TM, Kerns RD, Monson C, Scioli E. The development of an integrated treatment for veterans with comorbid chronic pain and posttraumatic stress disorder. Pain Med. 2009 Oct;10(7):1300-11. doi: 10.1111/j.1526-4637.2009.00715.x. PMID 19818040
- [Background] Kerns RD, Otis J, Rosenberg R, Reid MC. Veterans' reports of pain and associations with ratings of health, health-risk behaviors, affective distress, and use of the healthcare system. J Rehabil Res Dev. 2003 Sep-Oct;40(5):371-9. doi: 10.1682/jrrd.2003.09.0371. PMID 15080222
- [Background] Rakel BA, Blodgett NP, Zimmerman BM, Logsden-Sackett N, Clark C, Noiseux N, Callaghan J, Herr K, Geasland K, Yang X, Sluka KA. Predictors of postoperative movement and resting pain following total knee replacement. Pain. 2012 Nov;153(11):2192-2203. doi: 10.1016/j.pain.2012.06.021. Epub 2012 Jul 25. PMID 22840570
- [Background] Dindo L, Recober A, Marchman JN, Turvey C, O'Hara MW. One-day behavioral treatment for patients with comorbid depression and migraine: a pilot study. Behav Res Ther. 2012 Sep;50(9):537-43. doi: 10.1016/j.brat.2012.05.007. Epub 2012 May 27. PMID 22728646
- [Result] Dindo L, Zimmerman MB, Hadlandsmyth K, StMarie B, Embree J, Marchman J, Tripp-Reimer T, Rakel B. Acceptance and Commitment Therapy for Prevention of Chronic Postsurgical Pain and Opioid Use in At-Risk Veterans: A Pilot Randomized Controlled Study. J Pain. 2018 Oct;19(10):1211-1221. doi: 10.1016/j.jpain.2018.04.016. Epub 2018 May 17. PMID 29777950
- [Derived] Liu W, Dindo L, Hadlandsmyth K, Unick GJ, Zimmerman MB, St Marie B, Embree J, Tripp-Reimer T, Rakel B. Item Response Theory Analysis: PROMIS(R) Anxiety Form and Generalized Anxiety Disorder Scale. West J Nurs Res. 2022 Aug;44(8):765-772. doi: 10.1177/01939459211015985. Epub 2021 May 17. PMID 33998340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans indicated for orthopedic surgery and identified to be at-risk for poor outcomes were recruited following their indication clinic visit at the VAMC orthopedic clinic.
Pre-assignment Details: Eligible participants were randomized at their enrollment visit following phone screening. They were excluded if imminent risk of suicide. Active treatment groups received both ACT and TAU.
Groups:
- ACT + TAU: Acceptance and Commitment Therapy plus Treatment as Usual
- Treatment as Usual (TAU): Treatment as Usual
Period: Overall Study
Arm/Group | ACT + TAU | Treatment as Usual (TAU)
Started | 44 | 44
Completed | 40 | 35
Not Completed | 4 | 9
Not completed — Randomized but did not receive surgery | 4 | 8
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received surgery post randomization
Groups:
- Treatment as Usual: Treatment as usual - preoperative education and perioperative analgesia
- Total: Total of all reporting groups
Arm/Group | ACT + TAU | Treatment as Usual | Total
Number analyzed (Participants) | 40 | 34 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.1) | 63 (10.7) | 62.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 35 | 34 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 35 | 28 | 63
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 34 | 27 | 61
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 40 | 35 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percent of Veterans Willing and Able to Receive the ACT Intervention.
Description: The percent of veterans randomized to the ACT intervention who did receive the ACT intervention will be collected.
Time Frame: Enrollment to 3 months post surgery
Measure: Number; unit: percent
Arm/Group | ACT + TAU | Treatment as Usual (TAU)
Number analyzed (Participants) | 32 | 35
percent | 80 | 100

2. Primary Outcome: Amount of Pain Intensity on 0-10 Numeric Rating Scale
Description: Participants will be asked to rate the intensity of their maximum pain on a vertical, 0-10 numeric rating scale (0-10 NRS) with 0.5 increments at 3 months after surgery. Participants will be asked to provide a number that represents their highest pain intensity during the day if 0 is no pain and 10 is the most intense pain imaginable.
Time Frame: 3 months post surgery
Population: Intent-to-treat - with randomized participants who received surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ACT + TAU | Treatment as Usual
Number analyzed (Participants) | 40 | 35
score on a scale | 7.5 [5.5 to 8] | 8 [6 to 9]

3. Primary Outcome: Amount of Opioid Use
Description: Participants will be asked total daily dose of opioid medications at 3 months after surgery. All opioid doses converted to oral morphine equivalents.
Time Frame: 3 months post surgery
Population: Intent-to-treat - for participants who received surgery
Measure: Median (Full Range); unit: mg oral morphine
Groups:
- Treatment as Usual: Treatment as usual - preoperative education and peri-operative analgesia
Arm/Group | ACT + TAU | Treatment as Usual
Number analyzed (Participants) | 40 | 35
mg oral morphine | 0 [0 to 168] | 0 [0 to 200]

4. Primary Outcome: Length of Pain (Days)
Description: Participants will record their pain daily after surgery via an electronic (REDCap) or hardcopy log. When pain < 3 has been recorded for 5 consecutive days, the first date in the series will be used as the point of cessation and the length of time from surgery to this date will be calculated as the length of pain.
Time Frame: 6 months post surgery
Population: Intent-to-treat - with participants who received surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ACT + TAU | Treatment as Usual
Number analyzed (Participants) | 40 | 35
days | 66 [28 to 128] | 74 [32 to 184]

5. Primary Outcome: Length of Opioid Use (Days)
Description: Participants will record all pain medications (i.e. opioids and non-opioids) taken on a computerized pain medication form (or hardcopy log if participant does not have computer access available) until 3 months after surgery. The computerized pain medication form will list the drug name, route, dose, number taken, and date/time of each dose. When 0 doses of opioids have been recorded for 5 consecutive days, the first date in the series will be used as the point of cessation and the length of time from surgery to this date will be calculated as the length of opioid use.
Time Frame: 6 months post surgery
Population: Intent-to-treat - with participants who received surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ACT + TAU | Treatment as Usual
Number analyzed (Participants) | 40 | 35
days | 42.5 [30 to 96] | 51 [34 to 94]

ADVERSE EVENTS:
Arm/Group | ACT + TAU | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/34
Other Adverse Events (participants affected / at risk) | 2/40 | 6/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT + TAU (N=40) | Treatment as Usual (N=34)
Distress-based symptom increase (Psychiatric disorders) | 1 (1) | 5 (5) — Depression, anxiety, suicidal ideation
Pain increase (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No